CLINICAL TRIAL: NCT05399459
Title: Double-Blind, Randomized, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of Rimegepant for the Acute Treatment of Migraine in Japanese Subjects
Brief Title: Efficacy and Safety Study of Rimegepant for the Acute Treatment of Migraine in Japanese Subjects (Japan Only)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV3000-313; C4951022 (Other: Alias Study Number)
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Migraine
Keywords: Migraine; Headache; Acute Migraine
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Rimegepant 25 mg (Experimental): Single dose of 25 mg orally disintegrating tablet of rimegepant
  Interventions: Drug: Rimegepant 25 MG
- Rimegepant 75 mg (Experimental): Single dose of 75 mg orally disintegrating tablet of rimegepant
  Interventions: Drug: Rimegepant 75 MG
- Placebo (Placebo Comparator): Matching placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant 25 MG — Single dose of 25 mg orally disintegrating tablet of rimegepant
  Other Names: BHV3000
  Arms: Rimegepant 25 mg
Drug: Rimegepant 75 MG — Single dose of 75 mg orally disintegrating tablet of rimegepant
  Other Names: BHV3000
  Arms: Rimegepant 75 mg
Drug: Placebo — Matching placebo tablet
  Arms: Placebo

SUMMARY:
This study is being conducted to determine the appropriate dose of rimegepant in Japanese subjects, as well as to evaluate the efficacy, safety, and tolerability of rimegepant in Japanese subjects for the acute treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

Subject has at least 1 year history of migraines (with or without aura), consistent with a diagnosis according to the International Classification of Headache Disorder, 3rd Edition, including the following:

1. Migraine attacks present for more than 1 year with the age of onset prior to 50 years of age.
2. Migraine attacks, on average, lasting about 4-72 hours if untreated.
3. Not more than 8 attacks of moderate to severe intensity per month within the last 3 months.
4. Ability to distinguish migraine attacks from tension/cluster headaches.
5. Consistent migraine headaches of at least 2 migraine headache attacks of moderate or severe intensity in each of the 3 months prior to Screening Visit and maintains this requirement during the Screening period.
6. Less than 15 days with headache (migraine or non-migraine) per month in each of the 3 months prior to Screening Visit and maintains this requirement during the Screening Period.
7. Subjects on prophylactic migraine medication are permitted to remain on therapy if the dose has been stable for at least 3 months prior to the Screening Visit, and if the dose is not expected to change during the course of the study.
8. Subjects with contraindications for use of triptans may be included provided they meet all other study entry criteria.

Exclusion Criteria:

1. Subject has a history of migraine with brainstem aura (basilar migraine), hemiplegic migraine or retinal migraine.
2. History of use of analgesics (e.g. nonsteroidal anti-inflammatory drugs [NSAIDs] or acetaminophen) on ≥ 15 days per month during the 3 months (12 weeks) prior to the Screening Visit.
3. Subject history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Subjects with Myocardial Infarction (MI), Acute Coronary Syndrome (ACS), Percutaneous Coronary Intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months prior to screening.
4. Uncontrolled hypertension or uncontrolled diabetes (however subjects can be included who have stable hypertension and/or diabetes for at least 3 months prior to screening).
5. Subject with other pain syndromes, psychiatric conditions, dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, interfere with study assessments.
6. Subject has a history of gastric, or small intestinal surgery (including Gastric Bypass, Gastric Banding, Gastric Sleeve, Gastric Balloon, etc.), or has a disease that causes malabsorption.
7. The subject has a history or current evidence of any unstable medical conditions (e.g., history of congenital heart disease or arrhythmia, known or suspected infection, hepatitis B or C, or cancer) that, in the investigator's opinion, would expose them to undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course of the trial.
8. History of alcohol abuse and/or illicit drug use meeting DSM-V criteria for substance use disorder within 6 months of screening.
9. Participation in any other investigational clinical trial while participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 897 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- Japan (50):
  - Tokyo Dental College Ichikawa General Hospital, Ichikawa-shi, Chiba
  - Medical Corporation Seikokai Takanoko Hospital, Matsuyama, Ehime
  - Jinnouchi Neurosurgical Clinic, Kasuga-shi, Fukuoka
  - Ikeda Neurosurgical Clinic, Kasuga-shi, Fukuoka
  - SUBARU Health Insurance Society Ota Memorial Hospital, Ota-shi, Gunma
  - DOI CL Intern. Med./Neurol., Hiroshima, Hiroshima
  - Japanese Red Cross Asahikawa Hospital, Asahikawa-shi, Hokkaido
  - Higashi Sapporo Neurology and Neurosurgery Clinic, Sapporo, Hokkaido
  - Nakamura Memorial Hospital, Sapporo, Hokkaido
  - Konan Medical Center, Kobe, Hyōgo
  - Nishinomiya Municipal Central Hospital, Nishinomiya-shi, Hyōgo
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Kijima Neurosurgery Clinic, Kahoku-gun, Ishikawa-ken
  - Iwate Med. Univ. Uchimaru MC, Morioka, Iwate
  - Atsuchi Neurosurgery Hospital, Kagoshima, Kagoshima-ken
  - Tanaka Neurosurgical Clinic, Kagoshima, Kagoshima-ken
  - St. Marianna Univ. Hospital, Kawasaki-shi, Kanagawa
  - Fujitsu Clinic, Nakahara, Kanagawa
  - Atago Hospital, Kochi, Kochi
  - Umenotsuji Clinic, Kochi, Kochi
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Kyoto Okamoto Memorial Hospital, Kumiyama-cho, Kyoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Ishikawa Clinic, Sakyo-ku, Kyoto
  - Tatsuoka Neurology Clinic, Shimogyo-ku, Kyoto
  - Narikawa Neurological Clinic, Izumi-ku, Miyagi
  - Sendai Headache and Neurology Clinic, Medical Corporation, Sendai, Miyagi
  - Ooba CL Neurosurg. & Headache, Ōita, Oita Prefecture
  - Makabe Clinic, Okayama, Okayama-ken
  - Okayama City General Medical Center Okayama City Hospital, Okayama, Okayama-ken
  - Tominaga Clinic, Naniwa-ku, Osaka
  - Medical Research Institute KITANO HOSPITAL, PIIF Tazuke-kofukai, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Takase Intern. Med. Clinic, Toyonaka-shi, Osaka
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - JRC Shizuoka Hospital, Shizuoka, Shizuoka
  - Dokkyo Medical Univ. Hosp., Shimotsuga-gun, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokai university hachioji hospital, Hachioji-shi, Tokyo
  - Shinagawa Strings Clinic, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - USUDA CLINIC for internal medicine, Setagaya-ku, Tokyo
  - Tokyo Headache Clinic, Shibuya-Ku, Tokyo
  - Fukuuchi Pain Clinic, Shinjuku-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Nishiogi Pain Clinic, Suginami-ku, Tokyo
  - Suzuki Kei Yasuragi clinic, Tachikawa, Tokyo
  - Sakura Neuro Clinic, Toyama, Toyama
  - Nagamitsu Clinic, Hofu-shi, Yamaguchi
  - Nagaseki Headache Clinic, Kai-shi, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Ikeda K, Matsumori Y, Kudo M, Ishikawa T, Hoshino Y, Yoshimatsu H, Thiry A, Arakawa A, Croop R, Fullerton T, Sakai F, Takeshima T. Efficacy and safety of rimegepant for the acute treatment of migraine in Japan: A dose-ranging, double-blind, randomized controlled trial. Headache. 2025 Nov-Dec;65(10):1811-1820. doi: 10.1111/head.14994. Epub 2025 Jun 30. PMID 40586377
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-313

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 897 enrolled participants, 803 were randomized to receive study treatment.
Groups:
- Rimegepant 25 mg: Participants were randomized to receive orally disintegrated tablet (ODT) of rimegepant 25 milligram (mg) and of placebo (matched to rimegepant 75 mg) sublingually when they experienced a migraine headache of moderate to severe intensity, within 45 days of randomization on Day 1.
- Rimegepant 75 mg: Participants were randomized to receive ODT of rimegepant 75 mg and of placebo (matched to rimegepant 25 mg) sublingually when they experienced a migraine headache of moderate to severe intensity, within 45 days of randomization on Day 1.
- Placebo: Participants were randomized to receive ODT of placebo (each matched to rimegepant 25 and 75 mg) sublingually when they experienced a migraine headache of moderate to severe intensity, within 45 days of randomization on Day 1.
Period: Overall Study
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Started ((As randomized)) | 267 | 268 | 268 (One participant randomized in this group received rimegepant 25 mg.)
Efficacy Analysis Set (As Randomized) | 238 | 238 | 230 (One participant who was randomized to placebo received rimegepant 25 mg, included in this arm for efficacy analysis set.)
Safety Analysis Set (As Treated) | 239 (One participant who was randomized to placebo received rimegepant 25 mg, included in this arm for safety analysis set.) | 238 | 229
Completed ((As randomized)) | 237 | 238 | 230
Not Completed | 30 | 30 | 38
Not completed — Randomized but not treated | 29 | 30 | 38
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of participants in the enrolled analysis set (participants who signed an informed consent form and were assigned a participant identification number) and who had taken the study drug (rimegepant 25 mg, rimegepant 75 mg, or placebo). One participant who was randomized to the placebo group received rimegepant 25 mg. This participant in safety analysis set was included in rimegepant 25 mg arm and not in placebo arm.
Groups:
- Rimegepant 25 mg: Participants were randomized to receive ODT of rimegepant 25 mg and of placebo (matched to rimegepant 75 mg) sublingually when they experienced a migraine headache of moderate to severe intensity, within 45 days of randomization on Day 1.
- Total: Total of all reporting groups
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo | Total
Number analyzed (Participants) | 239 | 238 | 229 | 706
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (10.49) | 40.5 (11.25) | 41.4 (11.25) | 40.8 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 189 | 173 | 550
  Male | 51 | 49 | 56 | 156
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had Freedom From Pain at 2 Hours Post-Dose
Description: Pain freedom at 2 hours post-dose was defined as having a pain intensity of none at that time point. Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. Participants with score of 0 (no pain) were considered to have freedom from pain. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in Statistical Analysis Plan (SAP).
Time Frame: 2 hours post-dose
Population: Efficacy analysis set consisted of all participants in the full analysis set who were randomized only once, took the study drug, had a migraine of moderate or severe pain intensity at the time of treatment, and had post-dose efficacy data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 238 | 238 | 230
Percentage of participants | 21.0 [15.8 to 26.2] | 32.4 [26.4 to 38.3] | 13.0 [8.7 to 17.4]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Mantel Haenszel; Adjusted percentage difference = 19.4, 95% CI 2-sided [12.0 to 26.8] — Adjusted percentage difference (rimegepant 75 mg - placebo) stratified by randomization stratum with Mantel-Haenszel weighting

2. Secondary Outcome: Percentage of Participants With Pain Relief at 2 Hours Post-Dose
Description: Pain relief at 2 hours post-dose was defined as a pain intensity of none or mild at that time point. Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 238 | 238 | 230
Percentage of participants | 66.8 [60.8 to 72.8] | 79.0 [73.8 to 84.2] | 56.5 [50.1 to 62.9]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Mantel Haenszel; Adjusted percentage difference = 22.7, 95% CI 2-sided [14.5 to 30.9] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Who Had Freedom From Most Bothersome Symptom (MBS) at 2 Hours Post-Dose
Description: MBS freedom was defined as MBS reported before dosing that was absent post-dose. MBS included nausea, photophobia, or phonophobia. MBS were measured using a binary scale as 0= absent, 1= present. Participants who had score of 0 (MBS absent) were considered to have freedom from MBS. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 238 | 238 | 230
Percentage of participants | 53.4 [47.0 to 59.7] | 65.1 [59.1 to 71.2] | 50.4 [44.0 to 56.9]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.0011, Mantel Haenszel; Adjusted percentage difference = 14.8, 95% CI 2-sided [5.9 to 23.6] — Adjusted percentage difference (rimegepant 75 mg- placebo) stratified by randomization stratum with Mantel-Haenszel weighting

4. Secondary Outcome: Percentage of Participants With Ability to Function Normally at 2 Hours Post-Dose
Description: Functional disability was defined as a functional disability level of mildly impaired, severely impaired, or required bedrest. Participants rated the level of disability they perceived as a result of their migraine in performing normal actions using following level of severity: normal function, mild impairment, severe impairment, or required bedrest. Percentage of participants with a response of "normal function" at the 2 hours post-dose were reported in this outcome measure. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: 2 hours post-dose
Population: Efficacy analysis set consisted of all participants in the full analysis set who were randomized only once, took the study drug, had a migraine of moderate or severe pain intensity at the time of treatment, and had post-dose efficacy data. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 236 | 231 | 223
Percentage of participants | 36.0 [29.9 to 42.1] | 45.5 [39.0 to 51.9] | 26.9 [21.1 to 32.7]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Mantel Haenszel; Adjusted percentage difference = 18.8, 95% CI 2-sided [10.1 to 27.4] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 to 24 Hours Post-Dose
Description: Sustained Pain relief from 2 to 24 hours post-dose was defined as a pain intensity of none or mild at all time points from 2 to 24 hours post-dose. Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. Participants with score of 0 (with no pain) through 2 to 24 hours post-dose were considered to have sustained pain relief. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: 2 to 24 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 238 | 238 | 230
Percentage of participants | 48.3 [42.0 to 54.7] | 63.4 [57.3 to 69.6] | 31.7 [25.7 to 37.8]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Mantel Haenszel; Adjusted percentage difference = 31.7, 95% CI 2-sided [23.2 to 40.3] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Percentage of Participants Who Used Rescue Medication Within 24 Hours Post-Dose
Description: Percentage of participants who used rescue medications within 24 hours of administration of study drug were reported in this outcome measure. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: Within 24 hours post-dose
Population: Efficacy analysis set consisted of all participants in the full analysis set who were randomized only once, took study drug, had migraine of moderate or severe pain intensity at time of treatment and had post-dose efficacy data. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 238 | 238 | 229
Percentage of participants | 25.2 [19.7 to 30.7] | 19.7 [14.7 to 24.8] | 39.3 [33.0 to 45.6]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Mantel Haenszel; Adjusted percentage difference = -19.7, 95% CI 2-sided [-27.8 to -11.6] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Percentage of Participants With Sustained Pain Relief From 2 to 48 Hours Post-Dose
Description: Sustained pain relief from 2 to 48 hours post-dose was defined as a pain intensity of none or mild at all time points from 2 to 48 hours post-dose. Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. Participants with score of 0 (with no pain) through 2 to 48 hours post-dose were considered to have sustained pain relief. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: 2 to 48 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 238 | 238 | 230
Percentage of participants | 42.0 [35.7 to 48.3] | 60.5 [54.3 to 66.7] | 27.4 [21.6 to 33.2]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p < 0.0001, Mantel Haenszel; Adjusted percentage difference = 33.1, 95% CI 2-sided [24.7 to 41.6] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Percentage of Participants With Absence of Photophobia at 2 Hours Post-Dose
Description: Photophobia (sensitivity to light) status was measured as absent or present in the electronic diary (eDiary). Freedom from photophobia was defined as photophobia absent. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: 2 hours post-dose
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 162 | 159 | 153
Percentage of participants | 45.1 [37.4 to 52.7] | 59.1 [51.5 to 66.8] | 49.0 [41.1 to 56.9]
Statistical Analysis 1: Comparison: Rimegepant 75 mg vs Placebo; Test type: Superiority; p = 0.0707, Mantel Haenszel — P-value > 0.05; therefore, all secondary outcome measures listed after this outcome measure in the hierarchy were not tested; Adjusted percentage difference = 10.1, 95% CI 2-sided [-0.9 to 21.1] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 to 24 Hours Post-Dose
Description: Sustained pain freedom from 2 to 24 hours post-dose was defined as a pain intensity of none at all time points from 2 to 24 hours post-dose. Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. Participants with score of 0 (with no pain) through 2 to 24 hours post-dose were considered to have sustained pain freedom. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: 2 to 24 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 238 | 238 | 230
Percentage of participants | 13.9 [9.5 to 18.3] | 23.1 [17.8 to 28.5] | 6.5 [3.3 to 9.7]

10. Secondary Outcome: Percentage of Participants With Freedom of Phonophobia at 2 Hours Post-Dose
Description: Phonophobia (sensitivity to sound) status was measured as absent or present in the eDiary. Freedom from phonophobia was defined as phonophobia absent. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: 2 hours post-dose
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 131 | 108 | 108
Percentage of participants | 55.0 [46.4 to 63.5] | 66.7 [57.8 to 75.6] | 50.0 [40.6 to 59.4]

11. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom From 2 to 48 Hours Post-Dose
Description: Sustained pain freedom from 2 to 48 hours post-dose was defined as a pain intensity of none at all time points from 2 to 48 hours post-dose. Pain was measured on a 4-point Likert scale, with following scores: 0= none, 1= mild, 2= moderate, 3= severe. Participants with score of 0 (with no pain) through 2 to 48 hours post-dose were considered to have sustained pain freedom. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: 2 to 48 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 238 | 238 | 230
Percentage of participants | 11.8 [7.7 to 15.9] | 21.4 [16.2 to 26.6] | 6.1 [3.0 to 9.2]

12. Secondary Outcome: Percentage of Participants With Freedom From Nausea at 2 Hours Post Dose
Description: Nausea status was measured as absent or present in the eDiary. Freedom from nausea was defined as nausea absent. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: 2 hours post-dose
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 98 | 99 | 91
Percentage of participants | 68.4 [59.2 to 77.6] | 73.7 [65.1 to 82.4] | 62.6 [52.7 to 72.6]

13. Secondary Outcome: Percentage of Participants With Pain Relapse From 2 to 48 Hours Post-Dose
Description: Pain relapse from 2 to 48 hours post-dose was defined as pain intensity of mild, moderate, or severe at any time point post-dose after 2 hours post-dose for the subset of participants with pain intensity of none at 2 hours post-dose. Pain levels were assessed on a 4-point scale (none, mild, moderate, severe) using the eDiary. Formal statistical hypothesis testing was planned only for rimegepant 75 mg group with controlling type 1 error by the prespecified hierarchical gate-keeping procedure. For rimegepant 25 mg, no formal statistical hypothesis testing was conducted for any outcome measures as pre-specified in SAP.
Time Frame: 2 to 48 hours post-dose
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 50 | 77 | 30
Percentage of participants | 44.0 [30.2 to 57.8] | 33.8 [23.2 to 44.3] | 53.3 [35.5 to 71.2]

14. Secondary Outcome: Number of Participants With Adverse Events (AEs) by Intensity
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participants or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with the treatment. AE intensity included mild, moderate and severe. Mild AE is defined as AEs which is usually transient and may require only minimal treatment or therapeutic intervention. The event were not generally interfered with usual activities of daily living. Moderate AE is defined as AEs which is usually alleviated with additional specific therapeutic intervention. The event interfered with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the participants. Severe AE is defined as AE that interrupts with usual activities of daily living, significantly affects clinical status, or may require intensive therapeutic intervention.
Time Frame: From the day of signing informed consent up to end of treatment visit (approximately maximum up to 11 weeks)
Population: Safety analysis set consisted of participants in the enrolled analysis set who took the study drug (rimegepant 25 mg, rimegepant 75 mg, or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 239 | 238 | 229
Participants
  Mild | 16 | 19 | 12
  Moderate | 1 | 3 | 3
  Severe | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Serious AEs
Description: A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/ incapacity; resulted in congenital anomaly/birth defect in the off spring who received rimegepant were considered an important medical event.
Time Frame: From the day of signing informed consent up to end of treatment visit (approximately maximum up to 11 weeks)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 239 | 238 | 229
Participants | 0 | 1 | 0

16. Secondary Outcome: Number of Participants With Grade 3 to 4 Laboratory Test Abnormalities- Hematology
Description: Laboratory test abnormalities in hematology included: Eosinophils, Hemoglobin (high, low), Lymphocytes (high, low), Neutrophils, Platelets, White blood cell count (high, low). Laboratory abnormality events were graded according to National Cancer Institute Common Terminology Criteria For Adverse Events (NCI CTCAE) v5.0; grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death. Number of participants who had hematology parameter abnormality Grade 3 to 4 are reported in this outcome measure. Number of participants with non-zero laboratory abnormalities were reported in this outcome measure.
Time Frame: Baseline (Day 1) up to End of treatment visit (within 7 days of treatment) [approximately maximum up to 7 weeks]
Population: Safety analysis set consisted of participants in the enrolled analysis set who took the study drug (rimegepant 25 mg, rimegepant 75 mg, or placebo). Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 238 | 238 | 229
Participants | 1 | 0 | 0

17. Secondary Outcome: Number of Participants With Grade 3 to 4 Laboratory Test Abnormalities- Serum Chemistry
Description: Laboratory test abnormalities in serum chemistry included: alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, bicarbonate, Bilirubin (total), calcium (high, low), cholesterol (total), creatine kinase, creatinine, estimated glomerular filtration rate (eGFR), Modification of Diet in Renal Disease (MDRD), glucose, (high, low), lactate dehydrogenase low density lipoprotein (LDL) cholesterol (fasting, non-fasting), potassium (high, low), sodium (high, low), triglycerides (fasting, non-fasting), uric acid. Laboratory abnormality events were graded according to NCI CTCAE v5.0; grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death. Number of participants who had serum chemistry parameter abnormality Grade 3 to 4 are reported in this outcome measure. Number of participants with non-zero laboratory abnormalities are reported in this outcome measure.
Time Frame: Baseline (Day 1) up to End of treatment visit (within 7 days of treatment) [approximately maximum up to 7 weeks]
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 238 | 238 | 229
Participants
  Creatine kinase | 2 | 0 | 0
  LDL cholesterol | 4 | 3 | 4
  Triglycerides | 1 | 0 | 1

18. Secondary Outcome: Number of Participants With Grade 3 to 4 Laboratory Test Abnormalities- Urinalysis
Description: Laboratory test abnormalities in urinalysis included: Urine glucose, Urine protein, pH, specific gravity, ketones, nitrites, urobilinogen, leukocyte esterase, blood. If blood, protein or leukocytes are positive and determined clinically significant by the investigator, then the participants were returned for an unscheduled visit for microscopic examination. Laboratory abnormality events were graded according to NCI CTCAE v5.0; grade 1=mild, grade 2=moderate, grade 3=severe, grade 4=life-threatening consequences and grade 5=death. Number of participants who had urinalysis parameter abnormality Grade 3 to 4 are reported in this outcome measure. Number of participants with non-zero laboratory abnormalities are reported in this outcome measure.
Time Frame: Baseline (Day 1) up to End of treatment visit (within 7 days of treatment) [approximately maximum up to 7 weeks]
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
Number analyzed (Participants) | 236 | 238 | 228
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From the day of signing informed consent up to end of treatment visit (approximately maximum up to 11 weeks)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set consisted of participants in the enrolled analysis set who took the study drug (rimegepant 25 mg, rimegepant 75 mg, or placebo).
Arm/Group | Rimegepant 25 mg | Rimegepant 75 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/239 | 0/238 | 0/229
Serious Adverse Events (participants affected / at risk) | 0/239 | 1/238 | 0/229
Other Adverse Events (participants affected / at risk) | 3/239 | 3/238 | 2/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant 25 mg (N=239) | Rimegepant 75 mg (N=238) | Placebo (N=229)
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant 25 mg (N=239) | Rimegepant 75 mg (N=238) | Placebo (N=229)
Nasopharyngitis (Infections and infestations) | 3 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT05399459/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT05399459/SAP_001.pdf